CLINICAL TRIAL: NCT00691678
Title: Pase II Study of Glucosamine With Chondroitin on Joint Symptoms Induced By Aromatase Inhibitors in Breast Cancer Patients
Brief Title: Glucosamine and Chondroitin for Aromatase Inhibitor Induced Joint Symptoms in Women With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dawn L. Hershman (Other)
Responsible Party: Sponsor-Investigator, Dawn L. Hershman, Associate Professor of Medicine & Epidemiology, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAC8748
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Results first posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer; Joint Pain
Keywords: breast cancer; aromatase inhibitor; supportive care
MeSH Terms: conditions — Breast Neoplasms; Arthralgia | interventions — Chondroitin; Chondroitin Sulfates; Glucosamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- chondroitin and glucosamine (Experimental): Postmenopausal breast cancer patients that have joint symptoms induced by aromatase inhibitors and are receiving chondroitin and glucosamine.
  Interventions: Drug: Chondroitin; Drug: Glucosamine

INTERVENTIONS:
Drug: Chondroitin — 400mg chondroitin three times a day (TID) for twenty-four weeks
  Other Names: Chondroitin sulfate
Drug: Glucosamine — 500mg glucosamine TID for twenty-four weeks
  Other Names: Glucosamine sulfate

SUMMARY:
Investigators are hoping to learn if glucosamine with chondroitin can help relieve joint pain/stiffness associated with aromatase inhibitors.

DETAILED DESCRIPTION:
Due to early detection and improved treatments, women with breast cancer are living longer. The increase in breast cancer survival is largely due to the benefits of hormonal therapy, such as tamoxifen and aromatase inhibitors (AIs), for the treatment of hormone-sensitive breast cancer. Recent clinical trials have demonstrated that AIs are more effective than tamoxifen at reducing breast cancer recurrences. However, breast cancer patients receiving AIs have a higher incidence of osteoporosis, bone fractures and musculoskeletal symptoms, particularly joint pain and stiffness. Musculoskeletal pain, which occurs in up to 50% of patients treated with AIs, often does not respond to conventional pain medications, may lead to noncompliance, may cause major disability, and may interfere with quality of life. Many women are unable to tolerate these life-saving drugs because of severe joint pain, therefore, safe and effective treatments that alleviate these symptoms are needed.

ELIGIBILITY:
Inclusion Criteria:

* Age >21 years.
* Postmenopausal status defined as cessation of menses for >1 year or follicle-stimulating hormone (FSH) >20 milli-international units per milliliter or bilateral oophorectomy.
* History of stage I, II or III hormone receptor-positive breast cancer, without metastatic disease.
* Currently taking a third-generation aromatase inhibitor for at least 3 months.
* Clinical symptoms of knee and/or hand joint pain and/or stiffness for at least 3 months prior to study entry.
* Ongoing musculoskeletal pain/stiffness in hand and/or knee joints (50 or higher on the 100 point global assessment VAS) that started or increased since initiating aromatase inhibitor therapy, and has been present for at least 3 months.
* Patients must agree to refrain from use of glucosamine and chondroitin from sources outside of this study.
* If taking bisphosphonates, on a stable dose for at least 3 months and tolerating the dose. Patients must agree to refrain from initiating bisphosphonate use during the course of the study, therefore it is recommended that routine bone density testing be performed prior to enrollment or after completing trial.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Hemoglobin A1c <8 within the last year.
* Signed informed consent.

Exclusion Criteria:

* Use of glucosamine or chondroitin within the past three (3) months.
* Concurrent medical/arthritic disease that could confound or interfere with evaluation of pain or efficacy.
* History of significant collateral ligament, anterior cruciate ligament or meniscal injury of the index joint requiring surgery or non-weight bearing (requiring use of crutches or cane) for more than 3 weeks (minor ligamentous injury prior to 6 months is not an exclusion).
* History of bone fracture or surgery of the afflicted knees and/or hands within 6 months prior to study entry.
* Uncontrolled diabetes mellitus, defined as Hemoglobin A1c level of > 8%.
* History of any illness that, in the opinion of the investigator, might confound the results of the study or pose additional risk to the patient.
* Allergy to, or history of significant clinical or laboratory adverse experience associated with acetaminophen, glucosamine or chondroitin sulfate.
* Allergy to shellfish.
* Inability to understand and complete study questionnaires including questions requiring a visual analog scale (VAS) response.
* Inability to understand the study procedures and/or give written informed consent.
* Alcohol use in excess of 3 mixed drinks/day.
* Corticosteroid treatment was used or administered.
* Aspirin (up to 325 mg/day) for cardiovascular reasons may be continued.
* Intra-articular injection of hyaluronic acid or congeners into the study joint within 12 months.
* Topical analgesics (e.g., capsaicin preparations) to the study joint, or any oral analgesics (e.g., opiates, tramadol; with the exception of ibuprofen and acetaminophen) within 2 weeks of baseline visit or during the study.
* Implementation of any other medical therapy for arthritis within one month prior to entry.
* Other medications, unrelated to the patient's joint pain/stiffness must have been used at a stable dosage for at least 1 month. In addition, it should be anticipated that the dose of the concomitant medication will be stable during the entire treatment period.
* Participation in another clinical study with an investigational agent within the last 4 weeks.
* Exposure to glucosamine within 3 months or chondroitin sulfate within 3 months of Baseline Visit.
* Initiation of physical therapy or muscle conditioning program within 2 months prior to study entry.
* Concurrent use of the following medications and dietary supplements.

  * Chronic therapy with tetracycline or tetracycline derivatives.
  * Other new complementary or alternative regimens for the treatment of osteoarthritis, including, but not limited to, acupuncture, topical creams, oral agents, and magnets.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-10; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Hershman, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 53 women were enrolled in this study at baseline, 16 dropped out before the week 24 assessment. in total, there were 39 evaluable participants.
Pre-assignment Details: Of the 16 participants that dropped out of the study, 5 did so because of the number of pills, 8 due to adverse events and uncontrolled pain, and 3 dropped out due to other life events. 40 participants completed the 12 week assessment; 27 participants completed the 24 week assessment.
Period: Overall Study
Arm/Group | Chondroitin and Glucosamine
Started | 53
Completed | 37
Not Completed | 16
Not completed — Adverse Event | 5
Not completed — life events, pain | 11

BASELINE CHARACTERISTICS:
Groups:
- Chondroitin and Glucosamine: Postmenopausal breast cancer patients that have joint symptoms induced by aromatase inhibitors and are receiving chondroitin and glucosamine.
  Chondroitin: 400mg chondroitin TID for twenty-four weeks
  Glucosamine: 500mg glucosamine TID for twenty-four weeks
Arm/Group | Chondroitin and Glucosamine
Number analyzed (Participants) | 53
Age, Customized [Count of Participants; unit: Participants]
  18 - 58 years | 23
  59 - 78 years | 24
  > or = 79 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 38
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Change in WOMAC Score
Description: This is to demonstrate improvement in knee and/or joint pain and/or stiffness. The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The sum of the scores for all three subscales gives a total WOMAC score which ranges from 0-96. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Time Frame: Baseline and 24 weeks
Population: At completion of the study, there were 39 evaluable subjects (this excludes participants who were not available for follow-up) out of the 53 enrolled.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Chondroitin and Glucosamine
Number analyzed (Participants) | 39
Score on a scale | 24.9 (21.4)
Statistical Analysis 1: Comparison: Chondroitin and Glucosamine; This statistical analysis measures whether there is a statistically significant change, at the 5% significance level, between the mean WOMAC score among study participants at baseline and at week 24; Test type: Superiority; p = 0.004, t-test, 2 sided; Mean Difference (Final Values) = -13.3

ADVERSE EVENTS:
Time Frame: Up to 24 weeks
Arm/Group | Chondroitin and Glucosamine
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 51/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chondroitin and Glucosamine (N=53)
Nausea (Gastrointestinal disorders) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Flatulence (Gastrointestinal disorders) | 3 (3)
Heartburn (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Hiccough (Gastrointestinal disorders) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 1 (1)
Weight gain (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 14 (14)
Fatigue (Nervous system disorders) | 2 (2)
Allergic reaction (Immune system disorders) | 1 (1)
Bleeding at the biopsy site (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes